CLINICAL TRIAL: NCT07299331
Title: A Multicenter, Single-Arm, Prospective Clinical Study of Zanubrutinib, Rituximab, and Lenalidomide in the First-Line Treatment of Marginal Zone Lymphoma
Brief Title: Zanubrutinib, Rituximab, and Lenalidomide in the First-Line Treatment of Marginal Zone Lymphoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhengzhou University (Other)
Responsible Party: Principal Investigator, Mingzhi Zhang, Chief Physician, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-KY-1174-002
Record Dates: First submitted 2025-12-01; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-07

CONDITIONS: Marginal Zone Lymphoma(MZL)
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — zanubrutinib; Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Zanubrutinib, Rituximab, and Lenalidomide as the primary treatment for Marginal Zone Lymphoma (Experimental)
  Interventions: Drug: Zanubrutinib, Rituximab, and Lenalidomide as first-line treatment for Marginal Zone Lymphoma; Drug: Zanubrutinib, Rituximab, and Lenalidomide as the primary treatment for Marginal Zone Lymphoma

INTERVENTIONS:
Drug: Zanubrutinib, Rituximab, and Lenalidomide as first-line treatment for Marginal Zone Lymphoma — This study enrolls patients with marginal zone lymphoma who require the primary treatment. Participants receive a combined therapy consisting of zanubrutinib, rituximab, and lenalidomide.
Drug: Zanubrutinib, Rituximab, and Lenalidomide as the primary treatment for Marginal Zone Lymphoma — This study enrolls patients with marginal zone lymphoma who require the primary treatment. Participants receive a combined therapy consisting of zanubrutinib, rituximab, and lenalidomide.

SUMMARY:
The goal of this clinical trial is to learn if Zanubrutinib, Rituximab, and Lenalidomide works to treat marginal zone lymphoma as the first-line therapy. It will also learn about the safety of the treatment. The main questions it aims to answer are Does the combined therapy prolong patient survival? What medical problems do participants have when using this therapeutic approach? Researchers will observe the treatment to see if it works well than conventional therapies.

Participants will Administer drugs as required by the protocol Visit the clinic regularly for checkups and tests Keep a diary of their symptoms, examination and laboratory test indicators

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years
2. Histologically confirmed MZL in untreated stage III or IV and needed for therapy as determined by the treating physician
3. ECOG performance status 0-2
4. Expected survival ≥ 6 months
5. Adequate hematologic and organ function: absolute neutrophil count ≥1,000/mm3 (independent of growth factor support), platelet counts ≥75,000/mm3, serum aspartate transaminase or alanine transaminase less than 2.5 times the upper limit of normal (ULN), serum creatinine ≤1.5×ULN, and bilirubin ≤1.5×ULN unless bilirubin is due to Gilbert's syndrome, documented liver involvement with lymphoma, or of nonhepatic origin, in which case bilirubin should not exceed 3 g/dL, left ventricular ejection fraction (LVEF) of the heart≥ 50%
6. Women of childbearing potential and men who were sexually active were required to be practicing a highly effective method of birth control during and after the study
7. No history of other malignant tumors
8. At least one measurable lesion with a longest diameter of ≥ 1.5 cm or measurable lesions of extranodal lesions ≥ 1.0 cm.
9. Able to understand the study and provide signed Informed Consent Form

Exclusion Criteria:

1. Pregnant or lactating women
2. Active central nervous system lymphoma
3. Previous anti-tumor treatment
4. A severe immediate-type hypersensitivity reaction history for any of the drugs used in this study
5. History of stroke or intracranial hemorrhage within 6 months before study entry
6. Received a live attenuated vaccine within 4 weeks prior to enrollment History of human immunodeficiency virus, or active hepatitis C virus, or active hepatitis B virus infection, or any uncontrolled active systemic infection
7. Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any class 3 (moderate) or class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification
8. Other serious medical conditions that might have an impact on this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2031-04-30 (Estimated); Study Completion 2031-04-30 (Estimated)

PRIMARY OUTCOMES:
CRR | 2 years
  Complete remission rate

SECONDARY OUTCOMES:
ORR | 2 years
  Objective response rate
2 year-progress free survival rate | 2 years
  the time from the start of treatment to the time when the patient has progressed on the disease or dies due to any cause in 2 years.
TTR | From randomization up to 24 months post-randomization
  Time from randomization to the first documentation of Complete Response (CR) or Partial Response (PR) , verified by computed tomography (CT) and positron emission tomography (PET)-CT at least 6 weeks apart
DoR | From the date of first confirmed CR/PR up to 24 months post-confirmed response
  The interval from the date of first confirmed OR to the first evidence of progressive disease or death from any cause
OS | From randomization up to 24 months post-randomization
  The time from the date of randomization to the date of death from any cause
Incidence rate of adverse events | 2 years